CLINICAL TRIAL: NCT00174083
Title: Diagnosis of Active Tuberculosis in Endemic Area by Using Enzyme-Linked Immunospot Assay for Gamma-Interferon
Brief Title: Diagnosis of Active Tuberculosis by ELISPOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700717
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Tuberculosis
Keywords: Tuberculosis, TB-ELISPOT, active tuberculosis latent infection interferon
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Recent studies revealed that the ex vivo enzyme-linked immunospot (ELISPOT) assay for gamma interferon is a specific method for contact tracing of Mycobacterium tuberculosis infection. However, its use in endemic area and bacillus Calmette-Guérin (BCG)-vaccinated hosts has not been proved. We hypothesize that the TB-ELISPOT assay can be a rapid and accurate diagnostic tool for active tuberculosis in clinical suspects in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with fever or respiratory symptoms (cough, dyspnea, or hemoptysis) lasting for ≥ 2 weeks and have compatible radiographic findings were considered clinical suspects of TB.

Exclusion Criteria:

-

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2005-08; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Jann-Yuan Wang, MD, Principal Investigator — physician
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Wilkinson RJ, Vordermeier HM, Wilkinson KA, Sjolund A, Moreno C, Pasvol G, Ivanyi J. Peptide-specific T cell response to Mycobacterium tuberculosis: clinical spectrum, compartmentalization, and effect of chemotherapy. J Infect Dis. 1998 Sep;178(3):760-8. doi: 10.1086/515336. PMID 9728545
- [Background] Wilkinson KA, Wilkinson RJ, Pathan A, Ewer K, Prakash M, Klenerman P, Maskell N, Davies R, Pasvol G, Lalvani A. Ex vivo characterization of early secretory antigenic target 6-specific T cells at sites of active disease in pleural tuberculosis. Clin Infect Dis. 2005 Jan 1;40(1):184-7. doi: 10.1086/426139. Epub 2004 Dec 8. PMID 15614710
- [Background] Ulrichs T, Munk ME, Mollenkopf H, Behr-Perst S, Colangeli R, Gennaro ML, Kaufmann SH. Differential T cell responses to Mycobacterium tuberculosis ESAT6 in tuberculosis patients and healthy donors. Eur J Immunol. 1998 Dec;28(12):3949-58. doi: 10.1002/(SICI)1521-4141(199812)28:123.0.CO;2-4. PMID 9862331
- [Background] Ulrichs T, Anding R, Kaufmann SH, Munk ME. Numbers of IFN-gamma-producing cells against ESAT-6 increase in tuberculosis patients during chemotherapy. Int J Tuberc Lung Dis. 2000 Dec;4(12):1181-3. PMID 11144463
- [Background] Torres M, Herrera T, Villareal H, Rich EA, Sada E. Cytokine profiles for peripheral blood lymphocytes from patients with active pulmonary tuberculosis and healthy household contacts in response to the 30-kilodalton antigen of Mycobacterium tuberculosis. Infect Immun. 1998 Jan;66(1):176-80. doi: 10.1128/IAI.66.1.176-180.1998. PMID 9423855
- [Background] Skjot RL, Oettinger T, Rosenkrands I, Ravn P, Brock I, Jacobsen S, Andersen P. Comparative evaluation of low-molecular-mass proteins from Mycobacterium tuberculosis identifies members of the ESAT-6 family as immunodominant T-cell antigens. Infect Immun. 2000 Jan;68(1):214-20. doi: 10.1128/IAI.68.1.214-220.2000. PMID 10603390
- [Background] Schluger NW, Rom WN. The host immune response to tuberculosis. Am J Respir Crit Care Med. 1998 Mar;157(3 Pt 1):679-91. doi: 10.1164/ajrccm.157.3.9708002. No abstract available. PMID 9517576
- [Background] Richeldi L, Ewer K, Losi M, Bergamini BM, Roversi P, Deeks J, Fabbri LM, Lalvani A. T cell-based tracking of multidrug resistant tuberculosis infection after brief exposure. Am J Respir Crit Care Med. 2004 Aug 1;170(3):288-95. doi: 10.1164/rccm.200403-307OC. Epub 2004 May 6. PMID 15130907
- [Background] Ravn P, Demissie A, Eguale T, Wondwosson H, Lein D, Amoudy HA, Mustafa AS, Jensen AK, Holm A, Rosenkrands I, Oftung F, Olobo J, von Reyn F, Andersen P. Human T cell responses to the ESAT-6 antigen from Mycobacterium tuberculosis. J Infect Dis. 1999 Mar;179(3):637-45. doi: 10.1086/314640. PMID 9952370
- [Background] Pollock JM, Andersen P. The potential of the ESAT-6 antigen secreted by virulent mycobacteria for specific diagnosis of tuberculosis. J Infect Dis. 1997 May;175(5):1251-4. doi: 10.1086/593686. PMID 9129098